CLINICAL TRIAL: NCT05367583
Title: Cohort Study Assessing the Treatment Strategy for High-Risk Myelodysplastic
Brief Title: Cohort Study Assessing the Treatment Strategy for High-Risk Myelodysplastic Syndromes in Patients Under 70
Acronym: COMYRE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2012/22
Record Dates: First submitted 2019-07-02; First posted 2022-05-10 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic syndromes; Allogeneic Stem Cell Transplantation
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Allogeneic Stem Cell Transplantation — Allogeneic Stem Cell Transplantation

SUMMARY:
Myelodysplastic syndromes (MDS) are bone marrow malignant diseases resulting in ineffective haematopoiesis and subsequently, blood cell count decrease. Patients have anaemia responsible of fatigue and high heart frequency, thrombocytopenia responsible of increased risk of bleeding and neutropenia responsible of increased risk of infection. The patients suffering from MDS also are at increased risk of developing acute myeloblastic leukemia (AML). Allogeneic stem cell transplantation (alloSCT) remains the only curative option for patients with aggressive MDS. However, these patients are frequently ineligible for this kind of treatment, because of, for instance, age and co-morbidities. Thus, other treatment options are needed and Azacytidine (AZA), a hypomethylating agent is then proposed. With this COMYRE observatory study, we wanted to analyse which patients undergo alloSCT, why they are not eligible to alloSCT if it is the case, the overall survival of all the patients and if there are some factors which can influence this survival. It could help us to better identify the best candidate for alloSCT and those for other treatments such as AZA.

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) are a heterogeneous group of myeloid disorders due to qualitative defects of the hematopoietic stem cell, resulting in uneffective hematopoiesis, dysplasia of one or more lineages, and subsequently, various cytopenias. The patients suffering from MDS are at increased risk of developing acute myeloblastic leukemia (AML). Allogeneic stem cell transplantation (alloSCT) remains the only curative option for patients with intermediate-2 or high risk MDS according to International Prognostic Scoring System (IPSS). However, since these patients are frequently ineligible for this kind of treatment, because of age and co-morbidities, other treatment options were needed. Thank to AZA-001 trial results, Azacytidine (AZA), a hypomethylating agent is validated in Europe for the treatment of MDS patients who are not candidate for alloSCT. In most of cases, AZA is a well-tolerated drug comparing to more classical chemotherapy or alloSCT. Indeed, the most frequent reported side effects are fatigue, constipation, joints and muscle pains, cytopenias and these side effects rarely have significant clinical consequences. On the contrary, during alloSCT procedure, we could observe more infectious events, graft versus host disease, more toxicity.

In this COMYRE observatory study, all high risk MDS with age below 70 are included. The aim of the study is to analyse which patients undergo alloSCT and why they are not eligible to alloSCT if it is the case. We also want to analyse the overall survival of all included patients and we will try to identify if there are some factors which can influence this survival. Thus, it could help us to better identify the best candidate for alloSCT and those for other treatments such as AZA, regarding the benefit/toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old and <70 years old
* MDS-HR defined by an intermediate or high IPSS score (≥ 1.5), or IPSS revised ≥ to 4.5.
* Diagnosis affirmed by 2 myelograms at least 1 month apart or 1 single characteristic myelogram if prior haematological abnormalities on complete blood count present for more than 6 months
* Free informed consent signed by the patient and the investigator (at the latest on the day of inclusion and before any examination required by the study)
* Affiliate or beneficiary of a social security system

Exclusion Criteria:

* Age ≥ 70 years
* MDS-LR defined by a low IPSS score (<1.5), or revised IPSS <4.5
* Women of childbearing potential not using contraception, pregnant or breastfeeding
* Not affiliated to the Social Security system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MDS-HR defined by an intermediate or high IPSS score (≥ 1.5), or IPSS revised ≥ to 4.5
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2021-10-09 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient treated with Allogeneic stem cell transplantation (alloSCT) among enrolled patients | 3 months from baseline

SECONDARY OUTCOMES:
Evaluate the feasibility of the alloSCT: Proportion of patients with a donor | 3 months from baseline
Evaluate the effectiveness of iron chelation by measuring plasma ferritin (PF) (PF ≤ 1000 µg/L or PF > 1000 µg/L | Baseline and before alloSCT or 1 year from baseline for patient not treated with alloSCT
Evaluate the overall survival of patient treated and not treated with alloSCT | Until 5 year from baseline
Evaluate overall survival prognostic factors of patient treated and not treated with alloSCT | Baseline
Evaluate response rate to alloSCT or chemotherapy | Until 5 years from baseline
Evaluate toxicity to alloSCT (rate of systemic infection, rate of acute GVHD and rate of chronic GVHD) or chemotherapy (rate of systemic infection and rate of severe hemorrhage) | Until 5 years from baseline

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CH AGEN, Agen
  - Ch Bayonne, Bayonne
  - Chu de Bordeaux, Bordeaux
  - Institut Bergonie, Bordeaux
  - CH DAX, Dax
  - Ch Libourne, Libourne
  - Ch Marmande, Marmande
  - Ch Mont de Marsan, Mont-de-Marsan
  - CH PAU, Pau
  - Ch Villeneuve/Lot, Villeneuve-sur-Lot

IPD SHARING:
Plan to Share IPD: No